CLINICAL TRIAL: NCT03402672
Title: A Web-based E-health Application for Active Illicit Opioid Users Providing Information About Overdose and Infection Risk Factors and Encouraging HCV/HIV Testing and Medication Assisted Treatment Seeking
Brief Title: AWAITS: A Web-based E-health Application for Active Illicit Opioid Users
Acronym: AWAITS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Theresa Winhusen, PhD, Principal Investigator, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-1074-2
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Opioid-use Disorder; IV Drug Usage; Overdose; Drug Addiction; Substance Use Disorders
MeSH Terms: conditions — Opioid-Related Disorders; Drug Overdose; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AWAITS (Experimental): Participants who meet criteria will receive the AWAITS self-administered, e-health application intervention.
  Interventions: Other: self-administered, e-health application

INTERVENTIONS:
Other: self-administered, e-health application — AWAITS is a self-administered, e-health application and includes short videos in which patients who are successfully engaged in MAT discuss what they wish they had known about MAT when they were actively using. The intervention is designed to maximize "scalability" - the administration would entail handing an electronic device (e.g., tablet, laptop, etc.) to an individual who would then self-administer the intervention.

SUMMARY:
The purpose of this research study is to:

1. assess how participants like the AWAITS e-health application as measured by their feedback on the intervention
2. test the impact of AWAITS on knowledge about opioid overdose and risk-reduction strategies.
3. assess the proportion of participants who accept a list of local treatment providers
4. test the impact of AWAITS on interest in being tested for HCV/HIV.

DETAILED DESCRIPTION:
The pre-post study of AWAITS will: 1) assess the acceptability of AWAITS as measured by participant feedback about the intervention; 2) test the impact of AWAITS on knowledge about opioid overdose, as measured by the OOTAS; 3) assess the proportion of participants who accept a list of local MAT treatment providers; and 4) test the impact of AWAITS on interest in being tested for HCV/HIV.

The acceptability of AWAITS will be assessed with a feedback form which includes questions about how helpful the intervention was (scale of 1-4), what the patient liked most and least about the intervention, and any suggestions for improving it. The average (and standard deviation) for the rated helpfulness of the intervention will be derived and the qualitative data about what they liked most and least about the intervention and suggestions for improvement will be tabulated. Pre-/post-changes in the percent of correct knowledge assessment items (i.e., about overdose and MAT) and interest in HCV/HIV testing will be analyzed using a Wilcoxon signed-rank test. The proportion of participants accepting a list of local MAT treatment providers will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Not enrolled in MAT per self-report
3. Self-reports illicit opioid use

Exclusion Criteria:

3. Does not acknowledge reviewing "Information Sheet for Research" within REDCap

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-06-21 (Actual)

PRIMARY OUTCOMES:
3 sections of the OOTAS (signs of overdose, how to respond to an overdose, and MAT) | Day 1
  To test the impact of AWAITS on knowledge about opioid overdose

SECONDARY OUTCOMES:
Feedback on AWAITS | Day 1
  To assess the acceptability of the intervention
Acceptance of list of MAT providers | Day 1
  Assess relative interest in MAT post-AWAITS

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Winhusen, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Addiction Sciences Division, Cincinnati, Ohio, United States